CLINICAL TRIAL: NCT01144910
Title: A Prospective, Open Label, Single-center Study of the Long-term Prognosis of Moderate to Severe Bronchial Hyperresponsiveness (BHR) in Asthmatic Preschool Children.
Brief Title: The Long-term Prognosis of Moderate to Severe Bronchial Hyperresponsiveness (BHR) in Asthmatic Preschool Children
Acronym: BHR
Status: Withdrawn | Type: Observational
Why Stopped: Due to few capacities 2011 to 2016 the study was withdrawn.
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Schulze MD, Cosultant, Pediadric Allergy, Pulmonology and Cystic fibrosis, Johann Wolfgang Goethe University Hospital
Other Study IDs: KGU-317/09
Record Dates: First submitted 2010-06-01; First posted 2010-06-16 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Intrinsic Asthma; Allergic Asthma; Allergy; Bronchial Hyperresponsiveness
Keywords: asthma; preschool child; bronchial hyperresponsiveness; methacholine challenge test; atopy
MeSH Terms: conditions — Hypersensitivity; Bronchial Hyperreactivity; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BHR non-atopy: Patients from the outpatient Department of Allergy, Pneumology and Cystic fibrosis, children's hospital, Goethe-University, Frankfurt, Germany. Over a time-span of 5 years the investigators will explore the lung function and the bronchial hyperresponsiveness. Bronchial methacholine challenges will be performed at baseline and after 1, 3 and 5 years.
  Interventions: Other: methacholine challenge test
- BHR atopy: Patients from the outpatient Department of Allergy, Pneumology and Cystic fibrosis, children's hospital, Goethe-University, Frankfurt, Germany. Over a time-span of 5 years the investigators will explore the lung function and the bronchial hyperresponsiveness. Bronchial methacholine challenges will be performed at baseline and after 1, 3 and 5 years.
  Interventions: Other: methacholine challenge test

INTERVENTIONS:
Other: methacholine challenge test — 2 ml of liquid-dissolved methacholine in concentration of 16 mg/ml dosed in 5 steps of 0.01 mg, 0.1 mg, 0.4 mg, 0.8 mg, and 1.6 mg. 2 minutes after each step up an impulse oscillometry (IOS) and spirometry will be performed.
  the challenge will be stopped in case of a ≥ 20% decrease from baseline in FEV1 (PD20) and 0,2 mg Salbutamol will be given.
  Other Names: There are no other names
  Groups: BHR non-atopy
Other: methacholine challenge test — 2 ml of liquid-dissolved methacholine in concentration of 16 mg/ml dosed in 5 steps of 0.01 mg, 0.1 mg, 0.4 mg, 0.8 mg, and 1.6 mg. 2 minutes after each step up an impulse oscillometry (IOS) and spirometry will be performed.
  the challenge will be stopped in case of a ≥ 20% decrease from baseline in FEV1 (PD20) and 0,2 mg Salbutamol will be given.
  Other Names: There are no other names.
  Groups: BHR atopy

SUMMARY:
The aim of investigator´s clinical trial is to investigate 52 patients aged three to five years with viral-induced asthma and 52 patients aged three to five years with allergic asthma. Over a time-span of 5 years the investigators will explore lung function and bronchial responsiveness. The investigators plan to evaluate long-term clinical history of moderate to severe bronchial hyperresponsiveness in preschool children with asthma. Therefore factors like atopy in children, parental atopy and bronchial hyperresponsiveness will be explored.

DETAILED DESCRIPTION:
A positive family history with prevalence of atopy, eczema, wheezing are well-known factors predicting asthma. Caudri et al. found more important predictors like perinatal transmission, parental use of inhalative medications and wheezing/dyspnea out of viral infections(5). Measurement of BHR in children was in most studies a second outcome parameter.

Four visits will be performed, baseline and after 1, 3, and 5 years. At visit 1 the investigators will characterize all patients by a ISAAC survey. At each visit in children a methacholine challenge, a skin Prick test, eNO, RAST and total IgE will be performed. At visit 3 and 4 sputum will be induced. In parents only at the first visit a methacholine challenge will be performed. A genetic identification of ADAM33 gene from EDTA blood shall be provided. ADAMs are multidomain proteins with a metalloprotease domain, associated with airway remodelling. Visits should be kept in a time interval without asthma therapy and respiratory infection.

To examine the feasibility of methacholine challenges in preschool children data measured in 2006 will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age 3 to 6 years
* diagnosis asthma
* pulmonary function: FEV1 (% pred.)≥ 70%
* ability to carry out 2 reproducible flow volume loops
* moderate to severe BHR (PD20 FEV1 ≤ 0,3 mg methacholine)
* more than 4 weeks interval since last infection
* 8 hours washout period of Short Acting Beta Agonist
* 1 week washout period of Ipratropium Bromide
* 1 week washout period of Long Acting Beta Agonist
* 4 weeks washout period of Systemic Corticosteroids
* 4 weeks washout period of Leukotriene Antagonists

Exclusion Criteria:

* Age < 3 and > 6 Years
* Pulmonary function test: FEV1 (% pred.) < 70%
* Others chronic diseases or infections (e.g., HIV, tuberculosis, malignancy)
* Incapability to perform spirometry
* Current participation in another clinical trial

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients from the outpatient Department of Allergology, Pneumology and Cystic fibrosis, children's hospital, Goethe-University, Frankfurt, Germany
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change of severe bronchial hyperresponsiveness over time of five years. | five years
  Bronchial hyperresponsiveness will be defined by the provocation dose (PD) of methacholine causing a 20% drop of FEV1 (PD-20FEV1).

SECONDARY OUTCOMES:
Bronchial responsiveness of parents | two years
  In parents at first visit bronchial hyperresponsiveness will be defined by the provocation dose (PD) of methacholine causing a 20% drop of FEV1 (PD-20FEV1).
Impact of atopy | five years
  Influence of atopy on the time course of bronchial hyperresponsiveness.
eNO | five years
  Influence of the level of exhaled NO on the time course of BHR.
Total-IgE | five years
  Influence of the level of total-IgE on the time course of BHR

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schulze, Dr., Principal Investigator — Goethe University, Frankfurt, Germany
Locations (1):
- Goethe University, Frankfurt am Main, Germany

REFERENCES:
- [Background] Asher MI, Keil U, Anderson HR, Beasley R, Crane J, Martinez F, Mitchell EA, Pearce N, Sibbald B, Stewart AW, et al. International Study of Asthma and Allergies in Childhood (ISAAC): rationale and methods. Eur Respir J. 1995 Mar;8(3):483-91. doi: 10.1183/09031936.95.08030483. PMID 7789502
- [Background] Castro-Rodriguez JA, Holberg CJ, Wright AL, Martinez FD. A clinical index to define risk of asthma in young children with recurrent wheezing. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1403-6. doi: 10.1164/ajrccm.162.4.9912111. PMID 11029352
- [Background] Frank PI, Morris JA, Hazell ML, Linehan MF, Frank TL. Long term prognosis in preschool children with wheeze: longitudinal postal questionnaire study 1993-2004. BMJ. 2008 Jun 21;336(7658):1423-6. doi: 10.1136/bmj.39568.623750.BE. Epub 2008 Jun 16. PMID 18558639
- [Background] Matricardi PM, Illi S, Gruber C, Keil T, Nickel R, Wahn U, Lau S. Wheezing in childhood: incidence, longitudinal patterns and factors predicting persistence. Eur Respir J. 2008 Sep;32(3):585-92. doi: 10.1183/09031936.00066307. Epub 2008 May 14. PMID 18480107
- [Background] Caudri D, Wijga A, A Schipper CM, Hoekstra M, Postma DS, Koppelman GH, Brunekreef B, Smit HA, de Jongste JC. Predicting the long-term prognosis of children with symptoms suggestive of asthma at preschool age. J Allergy Clin Immunol. 2009 Nov;124(5):903-10.e1-7. doi: 10.1016/j.jaci.2009.06.045. Epub 2009 Aug 8. PMID 19665765
- [Background] Pijnenburg MW, Bakker EM, Hop WC, De Jongste JC. Titrating steroids on exhaled nitric oxide in children with asthma: a randomized controlled trial. Am J Respir Crit Care Med. 2005 Oct 1;172(7):831-6. doi: 10.1164/rccm.200503-458OC. Epub 2005 Jun 23. PMID 15976380
- [Background] Illi S, von Mutius E, Lau S, Niggemann B, Gruber C, Wahn U; Multicentre Allergy Study (MAS) group. Perennial allergen sensitisation early in life and chronic asthma in children: a birth cohort study. Lancet. 2006 Aug 26;368(9537):763-70. doi: 10.1016/S0140-6736(06)69286-6. PMID 16935687
- [Background] Nuijsink M, Hop WC, Sterk PJ, Duiverman EJ, de Jongste JC. Long-term asthma treatment guided by airway hyperresponsiveness in children: a randomised controlled trial. Eur Respir J. 2007 Sep;30(3):457-66. doi: 10.1183/09031936.00111806. Epub 2007 May 30. PMID 17537770
- [Background] Beydon N. Pulmonary function testing in young children. Paediatr Respir Rev. 2009 Dec;10(4):208-13. doi: 10.1016/j.prrv.2009.03.001. Epub 2009 Sep 25. PMID 19879511
- [Background] Beydon N. Assessment of bronchial responsiveness in preschool children. Paediatr Respir Rev. 2006;7 Suppl 1:S23-5. doi: 10.1016/j.prrv.2006.04.016. Epub 2006 Jun 5. PMID 16798575
- [Background] Holgate ST, Davies DE, Powell RM, Howarth PH, Haitchi HM, Holloway JW. Local genetic and environmental factors in asthma disease pathogenesis: chronicity and persistence mechanisms. Eur Respir J. 2007 Apr;29(4):793-803. doi: 10.1183/09031936.00087506. PMID 17400878
- [Background] Schulze J, Rosewich M, Riemer C, Dressler M, Rose MA, Zielen S. Methacholine challenge--comparison of an ATS protocol to a new rapid single concentration technique. Respir Med. 2009 Dec;103(12):1898-903. doi: 10.1016/j.rmed.2009.06.007. Epub 2009 Jul 10. PMID 19596563
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836
- [Background] Hagmolen of ten Have W, van den Berg NJ, van der Palen J, Bindels PJ, van Aalderen WM. Validation of a single concentration methacholine inhalation provocation test (SCIPT) in children. J Asthma. 2005 Jul-Aug;42(6):419-23. doi: 10.1081/JAS-67934. PMID 16293536